CLINICAL TRIAL: NCT04488159
Title: IMmunoscore Associated Decision GuIdance for AdjuvaNt Chemotherapy and Physical Exercise in Stage III Colon Cancer (iMAGINE): a Prospective, Randomized, Open-label, Multicenter, Phase III Clinical Trial
Brief Title: Immunoscore As Decision Guidance for Adjuvant Chemotherapy in Colon Cancer
Acronym: iMAGINE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Johannes Laengle, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Johannes Laengle, MD, PhD, Sponsor-Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iMAGINE; 2020-000401-91 (EudraCT Number)
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer Stage III
Keywords: Colon cancer; Immunoscore; CAPOX; FOLFOX; Physical exercise
MeSH Terms: conditions — Colonic Neoplasms; Motor Activity | interventions — Capecitabine; Oxaliplatin; Fluorouracil; Leucovorin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunoscore stratification (Experimental): * Immunoscore low (I-Low; I0-1): 3 months CAPOX (oxaliplatin 130 mg/m2 IV over 2 h and capecitabine 1000 mg/m2 PO twice daily (days 1-14). 21-day treatment cycle.). Concomitantly, standardised physical excise (stair walking excise twice a week for 12 weeks), which will be monitored by an electronic sports device.
  * Immunoscore intermediate-high (I-IntHi; I2-3): 6 months FOLFOX (oxaliplatin 85 mg/m2 IV (on day 1) and folinic acid 200 mg/m2 IV over 2 h, followed by a bolus of fluorouracil 400 mg/m2 IV over 2-4 min, followed by fluorouracil 600 mg/m2 IV over 22 h (for 2 consecutive days). 14-day treatment cycle.)
  * Immunoscore high (I high; I4): no adjuvant treatment.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Leucovorin; Device: Immunoscore® assay; Other: Physical exercise
- TNM stratification (Active Comparator): * TNM-based low-risk (pT1, pT2 or pT3 and pN1): 3 months CAPOX (oxaliplatin 130 mg/m2 IV over 2 h and capecitabine 1000 mg/m2 PO twice daily (days 1-14). 21-day treatment cycle.)
  * TNM-based high-risk (pT4 and/or pN2): 6 months FOLFOX (oxaliplatin 85 mg/m2 IV (on day 1) and folinic acid 200 mg/m2 IV over 2 h, followed by a bolus of fluorouracil 400 mg/m2 IV over 2-4 min, followed by fluorouracil 600 mg/m2 IV over 22 h (for 2 consecutive days). 14-day treatment cycle.)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Capecitabine — Tablet
Drug: Oxaliplatin — Infusion
Drug: Fluorouracil — Infusion
Drug: Leucovorin — Infusion
Device: Immunoscore® assay — Whole-slide tissue analysis of CD3+ and cytotoxic CD8+ T cells in the tumor and in the invasive margin
  Arms: Immunoscore stratification
Other: Physical exercise — Increasing stair walking exercise twice a week over 12 weeks total.
  Arms: Immunoscore stratification

SUMMARY:
The overall aim of this study is to prospectively validate the superiority of the Immunoscore as a decision guidance for adjuvant chemotherapy in stage III colon cancer patients, in comparison to the conventional TNM-based high- or low-risk classification.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* All sexes
* Histologically confirmed stage III carcinoma of the colon
* Medical need for an adjuvant chemotherapy
* Suitable to withstand the course of an adjuvant chemotherapy
* Written informed consent form (ICF) for participation in the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Neoadjuvant treatment
* Metastatic disease
* Pregnancy, breastfeeding or expectancy to conceive
* Disagreement of participants with reproductive potential to use contraception throughout the study period and for up to 180 days after the last dose of study therapy
* Uncontrolled or significant cardiovascular disease (myocardial infarction, uncontrolled angina, any history of clinically significant arrhythmias, QTc prolongation in males > 450 ms and > 470 ms in females, participants with history of myocarditis)
* Hepatitis B or C
* Human immunodeficiency virus (HIV)
* Immunodeficiency
* Allogeneic tissue or solid organ transplantation
* Systemic steroids or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Diagnosed and/or treated additional malignancy within 5 years of randomization, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin and/or curatively-resected in situ cervical and/or breast cancers
* Participants with serious or uncontrolled medical disorders
* Allergies and adverse drug reaction (history of allergy or hypersensitivity to study drug components, contraindications to any of the study drugs of the chemotherapy regimen)
* Other exclusion criteria: Prisoners or participants who are involuntarily incarcerated, participants who are compulsorily detained for treatment of either a psychiatric or physical (i.e. infectious disease) illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  Impact of Immunoscore stratification on DFS at 3 years (time from surgery to first observation of disease recurrence or death due to any cause)

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Impact of Immunoscore stratification on OS at 3 years (time from surgery to death due to any cause)
Time to recurrence (TTR) | 3 years
  Impact of Immunoscore stratification on TTR at 3 years (time from surgery to disease recurrence)
Treatment-related adverse events (AE) | 3 years
  Impact of Immunoscore stratification on treatment-related AEs assessed according to the latest Common Terminology Criteria of Adverse Events (CTCAE).
Health-related quality of life (HRQOL) | 3 years
  Impact of Immunoscore stratification on quality of life assessed by the latest version of the European Organization for Research and Treatment of Cancer (EORCT) Quality of Life Group (QLG) questionnaires C30 and CR29.
Cost analysis | 3 years
  Impact of Immunoscore stratification on treatment-related costs, assessed by cost-effectiveness analysis (CEA) according to the latest Good Research Practices for Cost-Effectiveness Analysis Alongside Clinical Trials of the International Society for Pharmacoeconomics and Outcomes Research (ISPOR).

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Galon, PhD, Principal Investigator — Laboratory of Integrative Cancer Immunology, INSERM, Cordeliers Research Center
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No